CLINICAL TRIAL: NCT05095610
Title: Clinical Effects of Intermitent Continuous Glucose Monitoring (Flash) in Adult Patients With Type 1 Diabetes in an Spanish Public Health System
Brief Title: Clinical Effects of Intermitent Continuous Glucose Monitoring in Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Castilla-La Mancha Health Service (Other)
Responsible Party: Sponsor
Other Study IDs: C-455
Record Dates: First submitted 2021-09-30; First posted 2021-10-27 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; intermitent continous glucose monitoring; Flash
MeSH Terms: conditions — Diabetes Mellitus, Type 1; photopsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Adult Type 1 Diabetes: All adult patients with type 1 diabetes previously followed in the DIACAM study (see bellow reference).
  Sastre J, Pinés PJ, Moreno J, Aguirre M, Blanco B, Calderón D, Herranz S, Roa C, Lopez J; Grupo de estudio DIACAM 1. Metabolic control and treatment patterns in patients with type 1 diabetes in Castilla-La Mancha: the DIAbetes tipo 1 in Castilla La Mancha study. Endocrinol Nutr. 2012 Nov;59(9):539-46. doi: 10.1016/j.endonu.2012.07.003.
  Interventions: Device: Flash

INTERVENTIONS:
Device: Flash — Use of the device FreeStyle Libre, only commercialized system for intermitent continuous glucose monitoring.
  Other Names: FreeStyle Libre; iCGM

SUMMARY:
Observational cross-sectional multicenter study about clinical effect of intermitent continuous glucose monitoring (Flash) in adult type 1 diabetes patients in an Spanish public health system.

DETAILED DESCRIPTION:
Observational cross-sectional multicenter study about clinical effect of intermitent continuous glucose monitoring (Flash) in adult type 1 diabetes patients in an Spanish public health system.

All clinical variables are gathered from chart review. Data analysis is conducted using SPSS statistic software. Results are presented as mean +/- SD values. A paired Student´s t-test or Wilconxon signed test were used fr the analysis differences. Comparison between proportions were analyzed using a chi-square test. A P value <0.05 was considered statistically significant.

The protocolo was apporved by the reference Castilla-La Mancha Public Health Service Ethic Commitee. All participants provided written consent.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Type 1 diabetes.
* Age >18 years.
* Patients previously followed in the DIACAM study.

Exclusion Criteria:

* Any other kinds of diabetes.

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients >18 years with type 1 diabetes and previously followed in the DIACAM study (see reference).
Sampling Method: Non-Probability Sample
Enrollment: 1121 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
HbA1c difference | 1 year
  Difference in HbA1c before initiating iCGM compared with HbA1c levels after one year of treatment.

SECONDARY OUTCOMES:
Frequency of SBGM | 1 year
  Daily number of blood capilary test fot glycemia determination.
Adherence to Flash | 1 year
  Time of use of Flash glucose monitoring (% possible time of use)
TIR | 1 year
  Time in range (TIR, 3.9-10 mmol/L) of the interstitial glucose
TAR | 1 year
  Time above range (TAR, >10 mmol/L) of the interstitial glucose
TBR | 1 year
  Time bellow range (TBR, <3.9 mmol/L) of the interstitial glucose
%CV | 1 year
  Percentage of the variation coefficient (%, >36% is considered high levels)
Body weight | 1 year
  Total corporal body weight (Kg)
Insulin dose | 1 year
  Daily insulin dose requirements (UI/Kg/d)

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - La Mancha- Centro Hospital, Alcázar de San Juan, Ciudad Real
  - Santa Barbara Hospital, Puertollano, Ciudad Real
  - Virgen de Altagracia Hospital, Valdepeñas, Ciudad Real
  - Virgen del Prado Hospital, Talavera de la Reina, Toledo
  - Albacete University Hospital, Albacete
  - Obispo Rafael Torija, St., Ciudad Real
  - Guadalajara University Hospital, Guadalajara
  - Toledo University Hospital, Toledo

IPD SHARING:
Plan to Share IPD: Undecided
After approval for the rest ot investigators.

REFERENCES:
- [Background] Sastre J, Pines PJ, Moreno J, Aguirre M, Blanco B, Calderon D, Herranz S, Roa C, Lopez J; Grupo de estudio DIACAM 1. Metabolic control and treatment patterns in patients with type 1 diabetes in Castilla-La Mancha: the DIAbetes tipo 1 in Castilla La Mancha study. Endocrinol Nutr. 2012 Nov;59(9):539-46. doi: 10.1016/j.endonu.2012.07.003. Epub 2012 Oct 4. English, Spanish. PMID 23039989
- [Derived] Moreno-Fernandez J, Sastre J, Pines P, Calderon-Vicente D, Gargallo J, Munoz-Rodriguez JR. To evaluate the use and clinical effect of intermittently scanned continuous glucose monitoring in adults with type 1 diabetes: Results of a multicentre study. Endocrinol Diabetes Nutr (Engl Ed). 2023 Apr;70(4):270-276. doi: 10.1016/j.endien.2023.03.013. PMID 37116972